CLINICAL TRIAL: NCT06346925
Title: Food Effects of Hexapopal Ethanolamine Tablets (Dosed 2 Hours After a High-fat Meal) in Healthy Subjects
Brief Title: Study of the Food Effects of Herombopag Olamine Tablets in Healthy Subjects.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR8735-116
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Adult Patients With Chronic Primary ITP; Adult Patients With SAA Who do Not Respond Well to Immunosuppressive Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): Take Herombopag Olamine Tablets 7.5mg 30min after high-fat meal in the first cycle. in the second cycle, take Herombopag Olamine Tablets 7.5mg on an empty stomach
  Interventions: Drug: Herombopag Olamine Tablets
- Treatment group B (Experimental): Take Herombopag Olamine Tablets 7.5mg 30min on an empty stomach in the first cycle. In the second cycle, take Herombopag Olamine Tablets 7.5mg 30min fter high-fat meal
  Interventions: Drug: Herombopag Olamine Tablets

INTERVENTIONS:
Drug: Herombopag Olamine Tablets — Three Herombopag Olamine Tablets is administered to healthy subjects.

SUMMARY:
This study was designed as a single-center, randomized, open, two-cycle, cross-over trial. It is planned to enroll 18 healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Male or female aged 18-45 at screening (both inclusive)
3. Body mass index (BMI) at 19.0~28.0 kg/m2 (including critical value)
4. Subjects who are considered to be generally healthy, based on an assessment of medical history, physical examination and clinical laboratory data, as judged by the Investigator
5. Subjects (including male subjects) are willing to have no birth plan and voluntarily adopt effective contraceptive measures and no sperm donation plan from 2 weeks before screening to 3 months after the last administration of the study drug, and ensure the use of one or more contraceptive methods during sexual life during this period

Exclusion Criteria:

1. People who have or are currently suffering from any clinically serious medical conditions such as circulatory, endocrine, neurological, digestive, respiratory, hematology, immunological, psychiatric and metabolic abnormalities within the previous year or any other disease that can interfere with the test results;.
2. People with a history of deep vein thrombosis or other thrombotic disorders.
3. Prolonged QTcF on 12-ECG at screening (450 ms > men and >470 ms) (corrected for Fridericia's formula or other clinically significant abnormalities determined by the clinician)。
4. Those who test positive for hepatitis B surface antigen, hepatitis C antibody, syphilis antibody, and HIV antibody
5. Those with a positive pregnancy test.
6. Allergies, such as those with a known history of allergy to two or more substances; or anyone allergic to Hydrazopag Ethanolamine tablets and their excipients.
7. Those who had undergone surgery within 4 weeks prior to screening, or who planned to undergo surgery during the study.
8. Has taken any prescription, over-the-counter, herbal or health product within 14 days prior to screening or dosing.
9. Those who participated in any clinical trial and used any investigational drug within 3 months prior to screening.
10. Blood donation (or blood loss) and blood donation (or blood loss) ≥400 mL within 3 months before screening, or receiving blood transfusion
11. Those who have special dietary requirements and cannot comply with the diet and corresponding regulations provided by the test.
12. Those who smoked an average of 5 or more cigarettes per day in the month prior to screening or could not stop using any tobacco products during the test period.
13. Those who consumed an average of more than 14 units of alcohol per week (1 unit of alcohol ≈360mL beer or 45mL spirits with 40% alcohol content or 150mL wine) in the three months before screening, or who could not abrol during the test period.
14. Positive alcohol test.
15. Those who have a history of drug abuse, drug dependence or positive urine drug screening within 3 months prior to screening.
16. Patients with a history of needle fainting or blood fainting, or those who cannot tolerate venous puncture blood collection.
17. People with difficulty swallowing tablets
18. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0hour to 120hours after the last dosing
AUC0-t | 0hour to 120hours after the last dosing
AUC0-∞ | 0hour to 120hours after the last dosing

SECONDARY OUTCOMES:
Tmax | 0hour to 120hours after the last dosing
t1/2 | 0hour to 120hours after the last dosing
CL/F | 0hour to 120hours after the last dosing
V/F | 0hour to 120hours after the last dosing
Incidence and severity of adverse events (AEs) | from screening to 120 hours after the last dosing

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical Uniersity, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided